CLINICAL TRIAL: NCT00926055
Title: Effects on Atherosclerosis Regression of Ezetimibe Monotherapy or Ezetimibe Plus Simvastatin Combination Therapy: Evaluation by Fluorodeoxyglucose Positron Emission Tomography
Brief Title: Effects on Atherosclerosis Regression of Ezetimibe or Ezetimibe Plus Simvastatin; Evaluated by Fluorodeoxyglucose Positron Emission Tomography (FDG-PET)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University (Other)
Responsible Party: Kyung Mook Choi, Korea University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01-2007-000-20546-0
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2010-06

CONDITIONS: Atherosclerosis
Keywords: high risk patients in atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Ezetimibe; Ezetimibe, Simvastatin Drug Combination; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention)
- Ezetimibe (Active Comparator)
  Interventions: Drug: Ezetrol (Ezetimibe)
- Ezetimibe/Simvastatin (Experimental)
  Interventions: Drug: Vytorin (Ezetimibe + Simvastatin)

INTERVENTIONS:
Drug: Ezetrol (Ezetimibe) — Ezetrol - 10 mg once daily for 3 months
  Arms: Ezetimibe
Drug: Vytorin (Ezetimibe + Simvastatin) — Vytorin - 10/20 mg once daily for 3 months
  Arms: Ezetimibe/Simvastatin

SUMMARY:
18F-fluorodeoxyglucose (FDG) positron emission tomography (PET) is a promising tool for identifying and quantifying vascular inflammation within atherosclerotic plaques. Therefore, in this study the investigators intend to compare the effect of ezetimibe monotherapy or ezetimibe plus statin combination therapy on the atherosclerosis regression using FDG-PET.

ELIGIBILITY:
Inclusion Criteria:

* hsCRP > 2 mg/L and LDL cholesterol > 130 mm/dL

Exclusion Criteria:

* history of cardiovascular disease
* diabetes
* uncontrolled hypertension
* active infection
* previous anti-hyperlipidemic agents within 6 months
* previous steroid or anti-inflammatory agents within 6 months
* liver disease
* renal disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
The difference of FDG uptake quantified by measuring the standardized uptake value (SUV) corrected for body weight according to the treatment groups | 3 months later

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro, Seoul, South Korea